CLINICAL TRIAL: NCT04811872
Title: Evaluation of the Effect of Placental Transfusion on Hemodynamics in Premature Newborns
Brief Title: Placental Transfusion Effect on Hemodynamics of Premature Newborns
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Marwa Mohamed Farag (Other)
Responsible Party: Sponsor-Investigator, Marwa Mohamed Farag, Primary Investigator and Lecturer in Pediatrics, Faculty of Medicine, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0106459
Record Dates: First submitted 2021-03-11; First posted 2021-03-23 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Pre-Term
MeSH Terms: conditions — Premature Birth | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intact umbilical cord milking (I-UCM) (Experimental)
  Interventions: Biological: Intact umbilical cord milking (I-UCM)
- Cut-umbilical cord milking(C-UCM) (Experimental)
  Interventions: Biological: Cut-umbilical cord milking(C-UCM)
- Delayed Cord Clamping (DCC ) (Experimental)
  Interventions: Biological: Delayed Cord Clamping (DCC)

INTERVENTIONS:
Biological: Intact umbilical cord milking (I-UCM) — Umblical cord milking will be performed by holding the newborn at or ∼20 cm below the level of the placenta. The cord will be pinched between 2 fingers as close to the placenta as possible and milked toward the infant over a 2-second duration. The cord will then be released and allowed to refill with blood for a brief 1- to 2-second pause between each milking motion. This will be repeated for 2-4 times. After completion, the cord will be clamped, and the neonate will be handed to the resuscitation team.
  Arms: Intact umbilical cord milking (I-UCM)
Biological: Cut-umbilical cord milking(C-UCM) — This technique involves clamping and cutting a long segment of the umbilical cord immediately at birth and passing the baby and the long cord to the pediatric provider, called C-UCM untwists the cord and milks the entire contents into the baby. Milking the cord 2-3 times before clamping may produce a similar placental transfusion as C-UCM.
  Arms: Cut-umbilical cord milking(C-UCM)
Biological: Delayed Cord Clamping (DCC) — Infants placed on the maternal abdomen or at the introitus below the level of placenta and waiting at least 30- to 60 seconds before clamping the cord.
  Arms: Delayed Cord Clamping (DCC )

SUMMARY:
The objective of this study is to perform ultrasound Doppler measurements to evaluate the hemodynamic changes associated with different methods of placental transfusion (Intact umbilical cord milking, cut- umbilical cord milking and delayed cord clamping) in premature neonates over the first days of life.

DETAILED DESCRIPTION:
This study will include a randomized controlled trial carried out on preterm neonates who will fulfill the eligibility criteria delivered at Alexandria University Children's Hospital. Evaluation of the outcome will be done only for those who admitted to the neonatal intensive care unit (NICU) at Alexandria University Children's Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Premature neonates ≤ 32 weeks gestational age regardless birth weight who will be admitted to neonatal intensive care unit in the first day of life.

Exclusion Criteria:

* Preterm babies >32 weeks
* Major congenital anomalies (complex cyanotic heart disease, major central nervous system anomalies).
* Evidence of head trauma causing major intracranial hemorrhage.
* Monochorionic multiples.
* Concern for abruptions, placenta previa or retroplacental hematoma.
* Cord accident, or avulsion at the time of delivery.
* Refusal to perform the intervention by the obstetrician

Ages: 0 Days to 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of superior vena cava flow (SVC) flow by echocardiography | up to 3 days of life
  Infants are placed in supine position on a flat surface and heart is imaged from a low subcostal view. SVC flow is identified by angling the beam anteriorly until the flow into the right atrium from SVC is seen using color Doppler. SVC diameter will be seen from a high parasternal long axis (PLAX) view. The transducer will be placed as close to the midline as possible to acquire directly anteroposterior views of SVC. Maximum and minimum internal diameters will be measured off-line from a frozen 2D image showing the vessel walls at the point where SVC starts to open into the right atrium. Due to the variation in vessel diameter through the cardiac cycle, mean of the maximum and minimum diameter is used for flow calculation. The velocity time integral (VTI) will be calculated from the Doppler velocity tracings and averaged over 5 consecutive cardiac cycles.
  SVC flow will be calculated using the Kluckow and Evans method = (VTI × 3.14 × (mean SVC diameter2/4) × heart rate) / body weight.
Measurement of fractional shortening (FS) by echocardiography | up to 3 days of life
  The FS is obtained from M-mode tracings or 2D imaging in the PLAX view at the tips of the mitral valve leaflets or in the parasternal short-axis (PSAX) view at the level of the papillary muscles. The left ventricular M-mode tracing is obtained from the PLAX or PSAX view. The cursor in M-mode should be placed perpendicular to the interventricular septum and posterior wall at the level of the posterior mitral valve leaflet. Left ventricular end-diastolic dimension (LVEDD) and left ventricular end-systolic dimension (LVESD) will be measured, and the FS is calculated using the following equation: FS (%) = (LVEDD - LVESD / LVEDD) × 100
Evaluation of ejection fraction (EF) by echocardiography | up to 3 days of life
  Left ventricular end-diastolic dimension (LVEDD) and left ventricular end-systolic dimension (LVESD) will be measured to calculate the ejection fraction.
  The EF is calculated using the following equation:
  EF (%) = (LVEDV - LVESV/ LVEDV)× 100
Evaluation of the pulse wave by echocardiography | up to 3 days of life
  The pulse wave (PW) Doppler across mitral inflow is composed of two waves: an E wave representing early passive ventricular filling (preload dependent) and an A wave representing late diastolic active filling as a result of atrial contraction.
Evaluation of left ventricular diastolic function by echocardiography | up to 3 days of life
  The mitral E/A ratio and velocity will be done for assessment of left ventricular diastolic function.
Evaluation of cardiac output (CO) | up to 3 days of life
  The echocardiographic assessment of the CO can be obtained by measuring cross-sectional area (CSA) of the left or RV outflow tract at the level of aortic or pulmonary annulus and by measuring the velocity time integral (VTI) at the level of aortic or pulmonary valve by pulsed wave Doppler, respectively. The CO is calculated by using the following equation:
  Cardiac Output (CO)=SV×HR= VTI× CSA× Heart Rate
Evaluation of patent ductus arteriosus (PDA) | up to 3 days of life
  The left-sided parasternal "ductal" view is the window to obtain a clear 2D image of the ductus arteriosus. The ultrasound probe is placed in a true sagittal plane to the left of the sternum with the marker pointing toward the head to obtain the ductal view. The PDA is visualized as a structure leaving the left side of the junction of the main pulmonary artery and the left pulmonary artery (LPA) toward the descending aorta. Color Doppler may be used to visualize the direction of transductal blood flow. The transdustal diameter will be measured in this view. Velocity and direction of the shunt during the cardiac cycle can be obtained by applying continuous wave.

CONTACTS AND LOCATIONS:
Locations (1):
- Neonatal Intensive Care Unit (NICU) of Alexandria University Maternity Hospital., Alexandria, Egypt

REFERENCES:
- [Derived] Farag MM, Thabet MAEH, Abd-Almohsen AM, Ibrahim HIAM. The effect of placental transfusion on hemodynamics in premature newborns: a randomized controlled trial. Eur J Pediatr. 2022 Dec;181(12):4121-4133. doi: 10.1007/s00431-022-04619-0. Epub 2022 Sep 21. PMID 36129535